CLINICAL TRIAL: NCT01009307
Title: San Francisco Bay Area Adult Glioma Prognosis Study Protocol
Brief Title: Study of Blood and Cheek Cell Samples From Patients With Glioma
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000437072; UCSF-H6539-04956-13A
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult brain stem glioma; adult giant cell glioblastoma; adult glioblastoma; recurrent adult brain tumor; adult gliosarcoma; adult mixed glioma; adult pineal gland astrocytoma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult pineoblastoma; adult pineocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma; Glioma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Pinealoma | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood and cheek cell samples from patients with glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine factors related to glioma survival in patients from two population-based case series collected in the San Francisco Bay Area between August 1991 and April 1994 (series 1) and May 1997 and August 1999 (series 2).

Secondary

* Determine vital status for 879 patients in the two San Francisco Bay Area population-based series through July 2004.
* Determine survival as a function of established, potential, and yet unstudied prognostic indicators.
* Gather data to validate results from this study with information from adult glioma patients enrolled prospectively at the UCSF-Neuro-Oncology clinic and through series 3 of the San Francisco Bay Area Adult Glioma Study; incorporate results from this study and other components of the SPORE into ongoing clinical investigations at the Brain Tumor Research Center and Neuro-Oncology Service at UCSF.
* Using funding from the organization Accelerate Brain Cancer Cure (ABC2), genotype several thousand single nucleotide polymorphisms (SNPs) from some study participants; assess these SNPs for potential relationship to glioma survival.

OUTLINE: Medical records of patients registered to the California Cancer Registry or the Northern California Cancer Center SEER are reviewed for mortality and treatment information related to the brain tumor. Blood and buccal specimens are collected from patients with newly diagnosed disease who are being seen at the UCSF Neuro-Oncology Service. The specimens are used for polymorphism and tumor marker studies and other pertinent data. Tumor specimens and treatment information related to the brain tumor are also collected from the SPORE Tissue Core.

Additional tumor makers are studied, including: chromosome 1p/19q, 7q studies; DNA repair and oxidative metabolism polymorphisms; and up to 2 tumor markers and 2 constitutive genotyping studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of glioma
* Meets 1 of the following criteria:

  * Participant in the Survival study of San Francisco Bay Area Adult Glioma Study (SFBAAGS) Series 1 and 2
  * Treated by UCSF Neuro-Oncology Service; diagnosed between Nov. 1, 2001 and June 30, 2006 and seen between Aug. 1, 2002 and June 30, 2006
  * Participant in SFBAAGS Series 3 (not seen at UCSF Neuro-Oncology Service) diagnosed between Nov. 1, 2001 and Oct. 31, 2004

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1709 (Actual)
Dates: Start 2001-10; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Factors related to glioma survival

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Wrensch, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States